CLINICAL TRIAL: NCT00705380
Title: Cognitive-Behavioral Treatment of Panic in Adolescence
Brief Title: Effectiveness of Cognitive Behavioral Therapy With Panic Control Treatment for Adolescents With Panic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sara Mattis, PhD, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R29MH058641 (NIH); R29MH058641 (NIH); DSIR CT-S
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive cognitive behavioral therapy with panic control treatment.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT) with panic control treatment (PCT) for adolescents
- 2 (Active Comparator): Participants will receive cognitive behavioral therapy with panic control treatment after a 12-week waitlist period.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT) with panic control treatment (PCT) for adolescents; Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) with panic control treatment (PCT) for adolescents — CBT with PCT treatment will consist of 11 weekly sessions that are designed to be developmentally appropriate for a younger population. The primary aim of this treatment will be to directly influence three aspects of panic attacks and general anxiety: the cognitive/misinterpretational aspect, the hyperventilatory response, and the conditioned reactions to physical sensations. Throughout treatment, participants will keep daily records of their anxiety and will complete self-monitoring forms to monitor panic attacks.
Behavioral: Waitlist control — During the 12-week waitlist period, participants will keep daily records of their anxiety and will complete self-monitoring forms to monitor panic attacks. Participants will also meet with a therapist every other week to discuss the nature of any panic attacks or address any concerns.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of cognitive behavioral therapy with a panic control treatment component in treating adolescents with panic disorder.

DETAILED DESCRIPTION:
More than 3 million people in the United States will experience a panic attack at some point in their lives. A panic attack occurs when a person experiences an intense feeling of sudden fear as well as physical sensations of breathlessness, rapid heart beat, and dizziness. Panic disorder, which is characterized by reoccurring panic attacks, often develops during childhood or adolescence and, if left untreated, can interfere with a child's normal development, relationships, school work, and psychological well-being. Cognitive behavioral therapy (CBT) with a panic control treatment (PCT) component is a type of psychotherapy that teaches new ways to control anxiety or panic attacks. It has been found to be effective in treating adults with panic disorder. However, more research is needed to determine if CBT with PCT, when adapted specifically for adolescents, is also effective in treating adolescents with panic disorder. This study will evaluate the effectiveness of CBT with a PCT component in treating adolescents with panic disorder.

Participation in this study will last up to 18 months. All participants will first undergo baseline assessments that will include a behavioral/psychological assessment while wearing a heart-rate monitoring device; questionnaires relating to experiences of anxiety, fear, and depression; and parent and child clinical interviews. Participants will then be assigned randomly to receive either immediate CBT with PCT or delayed CBT with PCT, which will occur after a 12-week waitlist period. CBT with PCT for all participants will include 11 weekly individual sessions, lasting 60 minutes each. During sessions, participants will learn specifically designed ways for adolescents to reduce or overcome panic attacks. Throughout treatment, participants will keep daily records of their anxiety and will complete self-monitoring forms to monitor panic attacks. During the 12-week waitlist period, the waitlist group participants will complete the same daily records and self-monitoring forms. The waitlist group participants will also meet with a therapist once every other week to discuss the nature of any panic attacks or address any concerns. Once all 12 weeks have passed, they will begin CBT with PCT. All participants will repeat the baseline assessments at Months 3, 6, and 12 after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for principal diagnosis of panic disorder or panic disorder with agoraphobia prior to treatment
* If on medication, must undergo a 1-month stabilization period for benzodiazepines or 3-month stabilization period for selective serotonin reuptake inhibitors or tricyclics before study entry

Exclusion Criteria:

* Positive diagnosis of schizophrenia, pervasive developmental disorder, organic brain syndrome, or mental retardation
* Current suicidal ideation
* Refusal of parent to accept random assignment to treatment condition
* Refusal of parent or adolescent to accept stabilization of medication

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 1998-07; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule-Child and Parent Versions: Clinical Severity Rating, Agoraphobia Ratings, Weekly Panic Attack Frequency Scores, and Monthly Panic Attack Frequency Scores | Measured at pretreatment; post-treatment; and Months 3, 6, and 12 of follow-up
Weekly Record of Anxiety and Depression (WRAD) | Measured at pretreatment; post-treatment; and Months 3, 6, and 12 of follow-up
The Panic Attack Record (PAR) | Measured at pretreatment; post-treatment; and Months 3, 6, and 12 of follow-up

SECONDARY OUTCOMES:
The Childhood Anxiety Sensitivity Index (CASI) | Measured at pretreatment; post-treatment; and Months 3, 6, and 12 of follow-up
Children's Depression Inventory (CDI) | Measured at pretreatment; post-treatment; and Months 3, 6, and 12 of follow-up
The Fear Survey Schedule for Children - Revised | Measured at pretreatment; post-treatment; and Months 3, 6, and 12 of follow-up
The Revised Children's Manifest Anxiety Scale | Measured at pretreatment; post-treatment; and Months 3, 6, and 12 of follow-up
Behavioral Approach Test (BAT) | Measured at pretreatment; post-treatment; and Months 3, 6, and 12 of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Mattis, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States